CLINICAL TRIAL: NCT02171091
Title: Impact of the Endotracheal Tube on Airway Inflammation: Prospective Analysis in Intubated ICU Patients
Brief Title: Intubated ICU Patients
Status: Terminated | Type: Observational
Why Stopped: Principal investigator leaving Washington University and halting studies
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201404106
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Patients Requiring Endotracheal Intubation
Keywords: endotracheal; intubation; airway; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and tracheal sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- study arm: One tracheal sample will be obtained using sterile (5 ml) sterile saline solution using irrigation and wall suction from each patient every day for 72 hours, total sampling time is approximately 10 seconds per specimen. Lung samples or fiberoptic obtained samples will be collected at same time intervals as the tracheal samples when possible and if they are done as standard of care. Samples will not be collected for research only and the time for this procedure will not be extended to collect extra tissue. A blood sample (10ml) will be collected simultaneously with the airway samples and also will be used for baseline control measurements.

SUMMARY:
The purpose of this research study is to determine how cell changes during endotracheal intubation and artificial lung ventilation affect lung inflammation.

Patients will undergo placement of an endotracheal tube (ETT) as standard of care. Tracheal (windpipe) lavage will be obtained each day for up to 72 hours. Lung samples or fiberoptic (lung) samples will be collected at the same time intervals when possible and if they are done as standard of care.

Blood samples will be obtained simultaneous with the collection of the trachael (windpipe) specimens.

ELIGIBILITY:
Inclusion Criteria

1. Ages 18 to 85
2. Required to have endotracheal intubation
3. Admitted to an intensive care unit

Exclusion Criteria

1. On immunosuppressive medications
2. Previous tracheal surgery
3. On azithromycin
4. Pregnancy
5. Cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients receiving endotracheal intubation in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Neutrophil changes | 72 hours
  Identifying indicators of neutrophil inflammatory changes that occur during 72 hours of tracheal injury secondary to endotracheal intubation.

SECONDARY OUTCOMES:
analyze neutrophil activation | 72 hours
  Analyze neutrophil activation in the distal airways in biological samples obtained simultaneously with tracheal samples and to correlate them with the development of lung inflammation.
correlate tracheal and lung neutrophil activation | 72 hours
  Correlate tracheal and lung neutrophil activation with development of pneumonia in ICU patients requiring mechanical ventilation.
determine the impact of airway (tracheal, lung) inflammation | 72 hours
  Determine the impact of airway (tracheal, lung) inflammation as determined by neutrophil activation on the length of stay (LOS), discharge, and readmission to ICU in the first 90 days post airway inflammation (VAP) diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Puyo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States